CLINICAL TRIAL: NCT03424954
Title: The Effect of a 30-day Automated Text Messaging Intervention on Hospital Based Acute Care Encounters Following Ileostomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB request IRB request
Sponsor: St. Louis University (Other)
Collaborators: Epharmix, Inc. (Industry)
Responsible Party: Principal Investigator, Grace Montenegro, MD, Assistant Professor, Department of Surgery, Division of General Surgery, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 28262
Record Dates: First submitted 2018-01-16; First posted 2018-02-07 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Ileostomy; Complications; Ileostomy - Stoma; Ileostomy Malfunction; Ileostomy Underactive; Complication of Surgical Procedure

STUDY DESIGN:
Intervention Model Description: All patients undergoing ileostomy surgery will receive the study intervention. We will compare to a historical control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EpxOstomy (Experimental): Post-operative ileostomy patients will receive the study intervention for 30 days following discharge from the hospital.
  Interventions: Behavioral: EpxOstomy

INTERVENTIONS:
Behavioral: EpxOstomy — A 30-day post-operative automated text-messaging intervention for home monitoring of ileostomy output

SUMMARY:
Each year a large number of patients undergo ileostomy surgery, a procedure in which a portion of the small intestine is attached to a hole in the abdominal wall, allowing for digested material to pass into a disposable bag worn attached to the skin. Ileostomies are performed for the treatment of a variety of diseases of the intestinal tract, such as inflammatory bowel disease, intestinal trauma, and gastrointestinal malignancy. Of the patients that undergo ileostomy surgery, 36% will require urgent medical care within the first 30 days of surgery. Most frequently, this is a result of dehydration due to excessive ostomy output. Thus, there is potential for significant improvement of the post-operative outcomes of ileostomy patients. Implementation of an automated text messaging system, EpxOstomy, can provide a way of monitoring patient's daily ostomy output and allow for timely intervention if output is outside normal limits, providing an effective way of improving patient outcomes while simultaneously reducing healthcare costs.

DETAILED DESCRIPTION:
Each year thousands of patients undergo ostomy surgery in the treatment of diseases such as colorectal cancer, Crohn's disease, diverticulitis, and ulcerative colitis. During the 30-day post-operative period, patients that undergo ileostomy have a 36.1% rate of acute healthcare encounter compared to 16.2% of patients undergoing similar surgery but with primary anastomosis. The 30-day hospital readmission rate for ileostomy patients due to dehydration and renal failure is 17%, with the median cost per colorectal surgery readmission being $8,885. Thus, there is substantial room for post-operative improvement in the care of ileostomy patients, both to reduce healthcare costs and improve patient quality of life. An automated text messaging system can provide a way to consistently monitor patients' ileostomy output, ensuring that patients are measuring their daily output as instructed and allowing for timely preemptive intervention should output be outside normal limits.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-90 years of age with phone or text receiving device access.
* English speaking
* Patients undergoing ileostomy surgery

Exclusion Criteria:

* Patients who do not have phone or text receiving device access
* Patients mentally unable to provide consent for the study
* Patients who do not speak English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Hospital-based acute health care encounters (HBAC) | 30 days following discharge
  The percentage of patients that require a HBAC (HBAC = readmissions + emergency department visits) due to post-op complications following ileostomy surgery. Medical records will be reviewed for readmissions or ED visits within 30-days following discharge. Additionally, the final message of the automated text-message intervention asks patients if they required readmission or ED care at any non-Saint Louis University Hospital facility(s).

SECONDARY OUTCOMES:
Patient response rates | throughout the 30 days of the intervention
  Automated message response data
Patient satisfaction survey results | One time, on day 30 of the intervention.
  Results of a patient survey administered via automated text-message after completion of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Montenegro, MD, Principal Investigator — Saint Louis University, Dept. of Surgery
Locations (1):
- SSM Health Saint Louis University Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan.

REFERENCES:
- [Background] Tyler JA, Fox JP, Dharmarajan S, Silviera ML, Hunt SR, Wise PE, Mutch MG. Acute health care resource utilization for ileostomy patients is higher than expected. Dis Colon Rectum. 2014 Dec;57(12):1412-20. doi: 10.1097/DCR.0000000000000246. PMID 25380008
- [Background] Paquette IM, Solan P, Rafferty JF, Ferguson MA, Davis BR. Readmission for dehydration or renal failure after ileostomy creation. Dis Colon Rectum. 2013 Aug;56(8):974-9. doi: 10.1097/DCR.0b013e31828d02ba. PMID 23838866
- [Background] Wick EC, Shore AD, Hirose K, Ibrahim AM, Gearhart SL, Efron J, Weiner JP, Makary MA. Readmission rates and cost following colorectal surgery. Dis Colon Rectum. 2011 Dec;54(12):1475-9. doi: 10.1097/DCR.0b013e31822ff8f0. PMID 22067174